CLINICAL TRIAL: NCT00071890
Title: Phase II/III Study Evaluating the Effect of IL-2 on Preservation of the CD4 T-Lymphocytes After Interruption of Anti-Retroviral TX in HIV Infected Patients With CD4 T-Lymphocyte Count Greater Than 500 Cells/mm(3) Who Have Received Anti-Retroviral TX
Brief Title: Phase II/III Study Evaluating the Effect of IL-2 on Preservation of the CD4 T-Lymphocytes After Interruption of Antiretroviral Treatment in HIV-Infected Patients With CD4 T-Lymphocyte Count Greater Than 500 Cells/mm3 Who Received Antiretroviral Tx
Acronym: ILIADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Irini Sereti, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040018; 04-I-0018 (Other: NIAID); ANRS 118 ILIADE (Other: ANRS)
Record Dates: First submitted 2003-11-03; First posted 2003-11-04 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: HIV Infections
Keywords: Interleukin 2; Treatment Interruption; HIV
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; aldesleukin; Antiretroviral Therapy, Highly Active; Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin 2 group (Active Comparator): HAART (standard of care) and three cycles of IL-2
  Interventions: Drug: Interleukin 2; Drug: HAART; Drug: Treatment interruption
- Control group (Active Comparator): HAART alone
  Interventions: Drug: HAART; Drug: Treatment interruption

INTERVENTIONS:
Drug: Interleukin 2 — Three cycles of IL-2 (6 MUI bid during 5 days = one cycle)
  Other Names: Interleukin-2; IL-2; aldesleukin
  Arms: Interleukin 2 group
Drug: HAART — HAART from week 0 to week 24
  Other Names: Antiretroviral treatment
Drug: Treatment interruption — HAART is interrupted from week 24 in both arms

SUMMARY:
This study will examine whether interleukin-2 (IL-2) given before the interruption of antiretroviral (ARV) treatment could significantly extend the period of time that a patient is temporarily not taking ARV treatment and also preserve CD4 counts above 350 cells per microliter. There will be an evaluation of the toxicity, or extremely harmful effects, of ARV, and the effect on quality of life.

The use of ARV medications has greatly improved the condition and mortality of HIV-infected patients. But when used long term, those medications have been associated with great toxicities and medication fatigue. As a result, patients may not adhere to ARV use, and resistance to viruses may grow. The CD4 molecule is on the surface of helper T-lymphocytes, or T-helper cells. It serves as the primary receptor for HIV-1 and HIV-2, allowing the virus to gain entry into its host. The CD4 count increases immediately in response to ARV, giving an estimate of the state of a patient's immune system. Thus, it is a strong marker of the immediate risk of an opportunistic infection, one that takes advantage of a person's weakened immune system. IL-2 is a molecule naturally produced by activated T cells. In patients with HIV, IL-2 treatment can increase CD4 counts but the clinical importance of this increase is not clear. This study will compare the decline in CD4 count, when ARV is interrupted, in two random groups of participants: (1) those who will receive three cycles of IL-2 (one every 8 weeks) in combination with ARV therapy for the first 24 weeks of the study before stopping ARV and (2) those who will receive ARV therapy without IL-2 for 24 weeks before stopping ARV.

Patients 18 years of age or older who have HIV-1 infection and who have been on ARV therapy for at least 1 year, and who currently have a CD4 count 500 cells per microliter or higher and never had a CD4 count of less than 200 cells per microliter and a viral load less than the limit of detection, may be eligible for this study.

Participants will undergo the following procedures and tests:

* Physical examination.
* Blood tests to measure blood lipids (fats), sugar, complete blood count including platelets, and chemistries.
* Assessment of fat distribution.
* Questionnaire about quality of life.

In addition, those participants who are randomly placed in the group receiving IL-2 and ARV will get an echocardiogram at the beginning of the study and at week 24. They will receive a starting dose of 6 million units of IL-2 as an injection under the skin twice a day. Each of the three IL-2 cycles will last 5 days. After the 24-week period, participants in both groups will stop taking ARV medications if their CD4 count is still equal to or greater than 500 cells per microliter. The study will continue into 120 weeks. Participants will be asked to continue to visit the clinic every 8 weeks for evaluation of their viral load and CD4 counts. Every 24 weeks, they will be asked to answer a questionnaire about their quality of life. Blood tests and other measurements will also be done as follow-up.

DETAILED DESCRIPTION:
The use of antiretroviral (ARV) medications has greatly improved morbidity and mortality of HIV-infected patients but long-term use of these agents has been associated with significant toxicities and medication fatigue that can lead to problems with adherence and eventual development of virologic resistance. The spectrum of ARV toxicities is broad including the development of lipodystrophy syndrome with lipid abnormalities and glucose intolerance or diabetes, while increasing evidence suggests an increased risk of cardiovascular complications in ARV-treated HIV-infected individuals. Current PHHS treatment guidelines recommend deferring ARV treatment initiation in asymptomatic HIV-infected individuals with CD4 count greater than or equal to 350 cells/micro liter, and treatment initiation after the CD4 count is less than 350 cells/micro liter. Several patients who started antiretroviral therapy at higher CD4 counts (based on older treatment initiation guidelines) or have experienced significant immunologic reconstitution after ARV initiation, elect to interrupt antiretroviral therapy until their CD4 count reaches the level of current recommendations for therapy initiation (less than 350 cells/micro liter).

Studies to date suggest that baseline and nadir CD4 count are the best predictors of a longer duration of treatment interruption that may be more beneficial with respect to reversal or delay of long-term ARV-associated toxicity and improved quality of life. It is known that intermittent cycles of IL-2 administration can lead to expansion of the CD4 pool and prolong survival of CD4 T cells. In this study the hypothesis tested is that IL-2 given prior to ARV treatment interruption could significantly prolong the period of ARV treatment interruption with preservation of CD4 counts above 350 cells/micro liter, and that this prolongation will be beneficial with respect to antiretroviral related toxicity and quality of life.

The study will have two parts: during the first part (24 weeks) patients will be randomized 1:1 to either receive three cycles or IL-2 with their ARV therapy or ARV therapy alone. In the second part (week 24 to week 120), all participants will interrupt therapy and restart when CD4 is less than 350 cells/micro liter. The main comparison will be at week 72, when the proportion of patients from the two groups who remain off drugs and have a CD4 greater than 350 cells/micro liter will be compared. At regular intervals (every 24 weeks) lipodystrophy measurements and quality of life questionnaires will be evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

HIV-1 infection confirmed by ELISA and Western Blot before screening.

Category A or B HIV-1 infection.

Antiretroviral treatment:

* started at least 12 months prior to screening visit;
* stable and continuous for at least 12 weeks prior to screening visit;
* modified no more than once for virologic failure.

IL-2 naive

CD-4(+) T-lymphocyte count greater than or equal to 500 cells/mm(3) in the twelve weeks prior to screening (historical) and at screening.

Nadir CD4(+) T-lymphocyte count greater than or equal to 200 cells/mm(3) prior to screening visit (that is, no measurement whose values may be less than 200/mm(3) since diagnosis of the HIV infection.

Plasma HIV RNA less than 50 copies/ml in the 12 weeks preceding screening (historical, less than limit of detection if different method and/or cut off used) and at screening.

For women of child-bearing age: use of effective contraception (hormonal such as birth control pill or injections, intrauterine device, surgical sterilization and/or mechanical barrier methods such as diaphragm or condoms); for all participants agreement to fully comply with prevention of transmission recommendations during periods of viremia if sexually active (latex condoms with or without additional barrier methods).

Desire to interrupt antiretroviral therapy.

Ability to sign informed consent (no later than W-2).

EXCLUSION CRITERIA:

Previous treatment with IL-2.

Combined treatment with interferon, other interleukins, anti-HIV vaccines, systemic (not topical or inhaled) corticosteroids and hydroxyurea within the previous 12 weeks.

Diagnosis of AIDS.

Acute infection in the 14 days preceding inclusion.

Pregnant, lactating woman desiring conception or not using contraception.

Hemoglobin less than 10 g/dl; neutrophils less than 1,000/mm(3); platelets less than 50,000/mm(3); creatinine greater than 1.5 times the upper limit of normal (N); bilirubin greater than 3N; AST or ALT greater than 3 N.

Progressive disease of malignant, psychiatric, cardiac, pulmonary, thyroid, renal or neurological (peripheral or central) origin or severe disorders of hemostasis.

Severe uncontrolled hypertension.

Previous or progressive pathology contraindicating the administration of IL-2.

History of extensive psoriasis, Crohn's disease or auto-immune disease involving severe complications.

HTLV-1 infection (ELISA positive).

Hepatitis B virus co-infection treated with lamivudine or tenofovir or adefovir.

Since atazanavir use can be associated with higher bilirubin levels (mostly indirect) in the absence of clinical consequences, subjects on atazanavir with bilirubin up to 4.5 times N may be allowed to participate if the levels have been stable and after approval by the PI or the PI designated covering physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Lévy, PHD, Study Chair — CHU Henri Mondor Créteil, FRANCE; Irini Sereti, MD, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Hospital Henri Mondor, Créteil, France

REFERENCES:
- [Background] Arno A, Ruiz L, Juan M, Jou A, Balague M, Zayat MK, Marfil S, Martinez-Picado J, Martinez MA, Romeu J, Pujol-Borrell R, Lane C, Clotet B. Efficacy of low-dose subcutaneous interleukin-2 to treat advanced human immunodeficiency virus type 1 in persons with </=250/microL CD4 T cells and undetectable plasma virus load. J Infect Dis. 1999 Jul;180(1):56-60. doi: 10.1086/314831. PMID 10353861
- [Background] Carr A, Emery S, Lloyd A, Hoy J, Garsia R, French M, Stewart G, Fyfe G, Cooper DA. Outpatient continuous intravenous interleukin-2 or subcutaneous, polyethylene glycol-modified interleukin-2 in human immunodeficiency virus-infected patients: a randomized, controlled, multicenter study. Australian IL-2 Study Group. J Infect Dis. 1998 Oct;178(4):992-9. doi: 10.1086/515653. PMID 9806026
- [Background] Carr A, Cooper DA. Adverse effects of antiretroviral therapy. Lancet. 2000 Oct 21;356(9239):1423-30. doi: 10.1016/S0140-6736(00)02854-3. PMID 11052597
- [Derived] Alexandre M, Prague M, Lhomme E, Lelievre JD, Wittkop L, Richert L, Levy Y, Thiebaut R. Definition of Virological Endpoints Improving the Design of HIV Cure Strategies Using Analytical Antiretroviral Treatment Interruption. Clin Infect Dis. 2024 Dec 17;79(6):1447-1457. doi: 10.1093/cid/ciae235. PMID 38819800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2003 to July 2006, 148 patients were randomized (81 in the IL-2 arm and 67 in the control arm in one centre of the NIH (USA) and 21 centres of the ANRS network (France).
Pre-assignment Details: 31 patients were not included because : CD4 below 500 (n=8), patient decision (n=6), HIV RNA < 50 copies/ml (n=5), neutropenia or high bilirubin(n=3), CD4 nadir below 200 (n=2),other diseases (n=2), AIDS (n=1), other reason (n=4)
Groups:
- Interleukin-2 Group: HAART and tree cycles of IL-2
- Control Group: HAART alone (without Interleukin-2)
Period: Overall Study
Arm/Group | Interleukin-2 Group | Control Group
Started | 81 (3 patients did not received Interleukin-2) | 67 (1 patients stopped HAART at week 0)
Completed | 81 (1 withdrawal 1 death 81 patients analysed) | 67 (1 withdrawal 1 lost of follow-up 1 death 67 patients analysed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interleukin-2 Group | Control Group | Total
Number analyzed (Participants) | 81 | 67 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 66 | 147
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (8) | 44 (9) | 43 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 66 | 54 | 120
Region of Enrollment [Number; unit: participants]
  France | 77 | 63 | 140
  United States | 4 | 4 | 8
CD4 at inclusion [Median (Inter-Quartile Range); unit: cells per mm3] | 770 [646 to 876] | 735 [625 to 834] | 747 [637 to 851]
CD4 nadir [Median (Inter-Quartile Range); unit: cells per mm3] | 326 [264 to 438] | 328 [259 to 355] | 326 [263 to 411]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without Failure of Strategy From Week 0 to Week 72
Description: A failure of strategy is defined on the first occurrence of one of the following events:
  * CD4 T-lymphocyte count becomes < 350 cells/mm3 between Wk0 and Wk72 (count confirmed by a 2nd measurement after 2-4 weeks
  * Planned interruption of therapy at Wk24 cannot be done for any reason;
  * Anti-retroviral treatment is restarted between Wk24 and Wk72 for any reason
  * Subject experiences clinical progression of HIV infection to a stage C AIDS diagnosis (appendix I)
  * Subject expires between Wk0 and Wk72 (whatever the cause of death)
  * Subject is lost to follow up
Time Frame: week 72
Population: Intent to treat analysis, missing = failure.
Measure: Number (95% Confidence Interval); unit: Pourcentage
Arm/Group | Interleukin-2 Group | Control Group
Number analyzed (Participants) | 81 | 67
Pourcentage | 73 [63 to 83] | 55 [43 to 67]
Statistical Analysis 1: Comparison: Interleukin-2 Group vs Control Group; Test type: Superiority or Other; p = 0.025, Chi-squared

2. Secondary Outcome: Changes in CD4 Counts at Week 72
Time Frame: week 72
Measure: Median (Inter-Quartile Range); unit: cells per mm3
Arm/Group | Interleukin-2 Group | Control Group
Number analyzed (Participants) | 81 | 67
cells per mm3 | 541 [398 to 702] | 453 [379 to 580]
Statistical Analysis 1: Comparison: Interleukin-2 Group vs Control Group; Test type: Superiority or Other; p = 0.069, Wilcoxon (Mann-Whitney) — Biphasic decline of CD4 after week 24 : first slope before W32 and weaker decline until W168.Slopes significantly different (all p values ≤0.0001) between the 2 groups, more pronounced in the IL-2 groups

3. Secondary Outcome: AIDS Events
Description: AIDS defined events according to CDC classification
Time Frame: Overall study
Population: * IL-2 arm : Oesophageal candidasis at W196
  * Control arm :Ocular B-cell lymphoma at W43,Oesophageal candidasis at W82, B-cell lymphoma at W104
Measure: Number; unit: event
Arm/Group | Interleukin-2 Group | Control Group
Number analyzed (Participants) | 81 | 67
event | 1 | 3

ADVERSE EVENTS:
Arm/Group | Interleukin-2 Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results with no delay specified